CLINICAL TRIAL: NCT01711255
Title: A Cross-Sectional Study of Coagulation in Multiple Sclerosis
Brief Title: Evaluation of Coagulation in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Bastyr University (Other)
Responsible Party: Sponsor
Other Study IDs: BU-12A-1323
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Coagulation; Alternative Medicine; Clotting; Complementary Medicine; Inflammation
MeSH Terms: conditions — Multiple Sclerosis; Thrombosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Six (6) whole blood vials of 10ml each will be collected from each subject. Three (3) will be stored for future use. Three will be used immediately for coagulation analysis using Sonoclot.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Subjects who have been diagnosed with clinically definite or probable multiple sclerosis as defined and recorded by board certified neurologist.
- Healthy controls: Adults age 18 and older who have not been diagnosed with any neurological, endocrine, or other chronic health condition. They must also be free of any recent acute illness that can impact inflammation/clotting.

SUMMARY:
Recent research in multiple sclerosis (MS) have suggested that altered coagulation and vascular inflammation may play a role in pathophysiology of MS. Sonoclot is viscoelastic method of analyzing clot formation. This instrument will be used to compare coagulation in individuals with MS to healthy controls. A 24-hour dietary recall and food frequency questionnaire will help determine whether coagulation is modified by fish consumption.

DETAILED DESCRIPTION:
This case-control study will recruit individuals with a diagnosis of MS and healthy controls. Individuals will be asked to come to Bastyr Clinical Research Center for a single study visit, at which time dietary intake, current medications and supplements, other medical diagnoses, and coagulation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically probable of clinically definite multiple sclerosis made by board certified neurologist. Subject must be willing to release medical information regarding diagnosis
* Controls must consider themselves healthy and be free of any neurological, autoimmune, endocrine or other chronic disease. Must also be free of any recent acute illness/injury that can influence inflammatory activity.
* Individuals must be 18 or older

Exclusion Criteria:

* Diagnosis of coagulation defect
* Use of anticoagulants (eg. warfarin, coumadin) or Aspirin within 30 days of entry.
* NSAID within 7 days of entry (dietary intake of fish oil or tumeric is acceptable)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be sixty (60) individuals with diagnosed or probable multiple sclerosis, verified by board certified neurologist, and forty (40) age and sex matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sonoclot Coagulation Spectrum (Sonoclot Signature) | Day 1
  The Sonoclot Coagulation Spectrum represents a combination of coagulation parameters, including activated clotting time, clot rate, time to peak, and peak amplitude. The mean value of all contributing parameters will be compared between cases and controls.

SECONDARY OUTCOMES:
ASA24 omega-3 fatty acid intake | 24 hour recall (24 hours prior to study visit)
  The ASA24, in combination with a medication history, will be used to evaluate whether omega-3 fatty acid intake is associated with reduced rates of coagulation in either cases or controls.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K Mischley, ND, Principal Investigator — Bastyr University - Clinical Research Center
Locations (1):
- Bastyr University Clinical Research Center, Kenmore, Washington, United States

REFERENCES:
- See also: Related info — http://www.bastyr.edu/research/clinical-research-center/integrative-neuroscience-research